CLINICAL TRIAL: NCT07116174
Title: A Prospective, Multi-center, Randomized Controlled Clinical Trial Evaluating the Effectiveness and Safety of Xcell Amnio MatrixTM (XAM) as Adjunct to Standard of Care (SOC) Therapy Compared to SOC Alone in the Management of Diabetic Foot Ulcers
Brief Title: A Prospective Clinical Study to Evaluate the Effectiveness and Safety of Xcell Amnio MatrixTM (XAM) in the Management of Chronic Non-healing DFUs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Horizon Medical Solutions (Network)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XAM-001
Record Dates: First submitted 2025-07-25; First posted 2025-08-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: DFU
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xcell Amnio MatrixTM (XAM) + Standard of Care (SOC) (Experimental)
  Interventions: Biological: Xcell Amnio Matrix
- Standard of Care (SOC) (Active Comparator)
  Interventions: Drug: Standard of Care (SOC)

INTERVENTIONS:
Biological: Xcell Amnio Matrix — A lyophilized amniotic membrane allograft
  Arms: Xcell Amnio MatrixTM (XAM) + Standard of Care (SOC)
Drug: Standard of Care (SOC) — The SOC will be based on investigator's choice
  Arms: Standard of Care (SOC)

SUMMARY:
The goal of this clinical trial is to evaluate the clinical outcomes of Diabetic Foot Ulcers (DFUs) treated with a weekly application of Xcell Amnio MatrixTM (XAM) as adjunct to standard of care (SOC) compared to SOC alone in male and female over the age of 18 years old. The main question it aims to answer is:

What is the proportion of subjects with complete wound closure during the 12 weeks of the treatment phase?

Participants:

* Will be screened and re-screened after 2 weeks to be assessed whether they meet the eligibility criteria
* Eligible subjects will receive study product application, and for 12 weeks will return to the clinic once every 7 days (±3 days) for treatment visits
* Subjects who complete the treatment will be followed up after 2 weeks

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL the following criteria at time of Screening:

1. Subject is 18 years of age or older.
2. Subject has diabetes mellitus (Type 1 or Type 2), requiring insulin or oral/injectable medications to control blood glucose levels
3. Glycosylated hemoglobin (HbA1c) level is <12%

   Note: Prior documented HbA1c within 12 weeks of Screening is acceptable.
4. Duration of ulcer is ≥ 4 weeks but ≤ 1 year, unresponsive to SOC
5. Ulcer area is ≥ 1.5cm2 and ≤ 20cm2 and with a clean, granulating base with minimal adherent slough at the Baseline Visit
6. Ulcer location is at or below the ankle (malleolus)
7. Subject is amenable to use of off-loading, as needed for planter ulcer
8. Ulcer extends through the full thickness of the skin but not down to muscle, tendon, or bone
9. Subject is at least 12 weeks post lower extremity revascularization procedure, if one has been performed.
10. Subject is in general good health, with no clinically significant medical conditions or abnormalities that, in the opinion of the Investigator, would interfere with study participation, the assessment of study endpoints, or pose additional risk to the subject.
11. Adequate circulation to the affected lower extremities as demonstrated by one of the following within 12 weeks of screening:

    1. Dorsum transcutaneous oxygen measurement (TCOM) ≥ 30 mmHg,
    2. Skin perfusion pressure (SPP) measurement ≥ 30 mmHg,
    3. Ankle-Brachial Index (ABI) ≥0.7 and ≤1.2, OR
    4. Toe-Brachial Index (TBI) ≥ 0.6
12. Subject is willing to use an acceptable method of contraception throughout the duration of the trial, if of childbearing potential.

    Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, patch, injectable, depot or vaginal) in conjunction with a barrier method (e.g., diaphragm, cervical cap, condom, spermicide or sponge), or female subject/partner's use of an implantable device (implantable rod or intrauterine device).

    Female subject/partners of non-childbearing potential are defined as surgically sterile (e.g., bilateral tubal ligation, hysterectomy) or two years postmenopausal at time of screening.

    All male subjects (excluding men who have been sterilized) with female partners of child-bearing potential must agree to consistently and correctly use a condom for the duration of the study. In addition, subjects may not donate sperm for the same time period.
13. Subject is able to read, understand and sign the informed consent form (ICF).
14. Subject is available and willing to complete all study assessments and can comply with standard of care (debridement, dressing changes etc.) as applicable.

Exclusion Criteria:

Subjects meeting ANY of the following criteria at time of Screening will be excluded from enrollment:

1. Clinical evidence of ongoing infection and/or receipt of IV, oral, or topical antimicrobials.
2. Wheelchair bound or bed-ridden (ambulatory with assistance is acceptable).
3. Ulceration at the site of amputation.
4. Undergoing renal dialysis.
5. Known or suspected malignancy in the target ulcer, or a history of cancer in the preceding 5 years (other than carcinoma in situ of the cervix or adequately treated non-melanoma skin cancer).
6. Documented history of osteomyelitis at the target ulcer location within 6 months of screening.
7. History of radiation at the ulcer site.
8. New York Heart Association Class III or IV congestive heart failure or uncontrolled cardiac dysrhythmia.
9. Diagnosis of autoimmune disease(s) (rheumatoid arthritis, lupus, psoriasis, Sjogren's syndrome) or arthritis requiring corticosteroid treatment.
10. Subject has received in the past 4 weeks or is scheduled to receive any of following medication or therapies during the course of the study:

    1. Immunosuppressants (including chronic systemic corticosteroids or application of topical steroids to the ulcer surface)
    2. Cytotoxic chemotherapy
    3. Growth hormone
    4. Oral or systemic antifungal or antituberculosis treatment
    5. Use of any investigational drug(s) or therapeutic device(s)
11. Target ulcer(s) previously treated with negative pressure, hyperbaric oxygen, or tissue engineered materials (e.g., Apligraf®, EpiFix® or Dermagraft®) or other scaffold materials (e.g., Oasis, Matristem) within 4 weeks prior to screening.
12. Target ulcer(s) anticipated to require negative pressure wound therapy or hyperbaric oxygen at any time during the study.
13. Healing of target ulcer is observed to be ≥35% at the end of the Run-in Period (between Screening and Baseline Visits)
14. Subject is pregnant or breastfeeding.
15. Presence of any other condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.
16. Active Charcot foot (stable chronic Charcot foot is not exclusionary).
17. Ulcers on toes 2, 3, 4, and/or 5 only (ulcer on plantar surface of the great toe only is not exclusionary).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with complete wound closure during the 12 weeks of the Treatment Phase | Baseline to12 weeks
  Complete wound closure is defined as 100% re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart.

SECONDARY OUTCOMES:
Wound Area Change (%) during the 12 weeks of the Treatment Phase | Baseline to 12 weeks
  Wound area change is defined as the percentage of wound area change as measured by SnapshotNIR wound imaging device.
Time to complete wound closure during the 12 weeks of the Treatment Phase | Baseline to 12 weeks
  The time of complete closure will be the visit when 100% re-epithelialization without drainage or dressing requirements was first achieved.
Change in pain in the target ulcer assessed using the Visual Analogue Scale (VAS) during the 12 weeks of the Treatment Phase. | Baseline to 12 weeks
  Minimum value: 0 Maximum value: 100 Higher scores indicate a better outcome (greater satisfaction or improved quality of life related to wound care).

OTHER OUTCOMES:
Change in quality of life using the WOUND-Q (patient-reported outcome measure) assessment | Baseline to 12 weeks
  Exploratory Outcome Measure Minimum value: 0 Maximum value: 100 Higher scores indicate a better outcome (greater satisfaction or improved quality of life related to wound care).
Changes in tissue perfusion (tissue oxygen saturation (StO2), oxyhemoglobin, and deoxyhemoglobin) as measured by SnapshotNIR wound imaging device. | Baseline to follow up visit at week 15
  Exploratory Outcome Measure
Incidence and severity of treatment-emergent adverse events (TEAEs) | Baseline to follow up visit at week 15
  Safety Outcome Measure
Incidence of withdrawals due to Adverse Events (AEs) | Baseline to follow up visit at week 15
  Safety Outcome Measure
Incidence of Treatment-Related Adverse Events | Baseline to follow up visit at week 15
  Safety Outcome Measure
Incidence of Serious Adverse Events (SAEs) | Baseline to follow up visit at week 15
  Safety Outcome Measure

CONTACTS AND LOCATIONS:
Locations (1):
- Richard C. Galperin, Dallas, Texas, United States